CLINICAL TRIAL: NCT02069665
Title: Assessing the Effectiveness of Integrative Treatment That Combines Interior and Exterior Treatment Plans in Pediatric Pneumonia: a Program by PRC National Clinical Research Base of Traditional Chinese Medicine for Major Diseases
Brief Title: Effectiveness Study of Integrative Treatment for Pediatric Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaoning University of Traditional Chinese Medicine (Other)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xuefeng Wang, Chief physician, Liaoning University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHLN-TCM-01
Record Dates: First submitted 2013-12-26; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Pneumonia
Keywords: pneumonia; pediatrics; viral
MeSH Terms: conditions — Pneumonia | interventions — Ribavirin; Guaifenesin; N-methylephedrine; Ibuprofen; Albuterol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Injection, medications and application (Experimental): Intravenous injection: Xiyanping injection, produced by Jiangxi Qing Feng Pharmaceutical Co., Ltd;
  Medications: according to TCM syndrome differentiations;
  * Wind-heat blocking lungs pattern (feng re bi fei zheng): Xiaoer Qingfei Heji (mixture), and Zhi Ke San (herbal powder to relieve cough)
  * Phlegm-heat blocking lungs pattern (tan re bi fei zheng): Xiaoer Qingfei Heji (mixture), and Hua Tan San (herbal powder to remove phlegm)
  External application: Fuxiong San
  Interventions: Other: Fuxiong San; Drug: Xiyanping injection; Drug: Xiaoer Qingfei Heji (mixture); Drug: Zhi Ke San; Drug: Hua Tan San
- Injection and medications (Active Comparator): Intravenous injection: Ribavirin Injection;
  Medications: symptomatic therapies
  * Guaifenesin Syrup, for removing phlegm, relieving gasp-cough;
  * Ibuprofen Suspension, and salbutamol in case of different symptoms
  Interventions: Drug: Ribavirin Injection; Drug: Guaifenesin Syrup; Drug: Ibuprofen Suspension; Drug: salbutamol

INTERVENTIONS:
Other: Fuxiong San — external application; 8-10cm wide, 0.3-0.5cm thick; 10mins for patient aged 1 to 3-year old; 15mins for those aged 3 to 5-year old; once daily
  Arms: Injection, medications and application
Drug: Xiyanping injection — ivd. 5 to 10 mg/(kg•d), plus 5% Glucose Injection, 80 to 100 ml, ivd. Once a day injection.
  Arms: Injection, medications and application
Drug: Ribavirin Injection — ivd. 10 to 20 mg/(kg•d), plus 5% Glucose Injection, 80 to 100 ml, ivd. Once a day injection.
  Arms: Injection and medications
Drug: Xiaoer Qingfei Heji (mixture) — children aged 6 months to 1 year old: 10 ml, orally taken three times daily; children aged 1 to 3 year old: 15 ml, orally taken three times daily; children aged 3 to 5 year old: 20 ml, orally taken three times daily;
  Arms: Injection, medications and application
Drug: Zhi Ke San — children aged 6 months to 1 year old: 0.5g, orally taken three times daily; children aged 1 to 3 year old: 1.5g, orally taken three times daily; children aged 3 to 5 year old: 2.0g, orally taken three times daily;
  Other Names: herbal powder to relieve cough
  Arms: Injection, medications and application
Drug: Hua Tan San — children aged 6 months to 1 year old: 0.5g, orally taken three times daily; children aged 1 to 3 year old: 1.5g, orally taken three times daily; children aged 3 to 5 year old: 2.0g, orally taken three times daily;
  Other Names: herbal powder to remove phlegm
  Arms: Injection, medications and application
Drug: Guaifenesin Syrup — children aged 6 months to 1 year old: 3ml, orally taken three times daily; children aged 1 to 3 year old: 5ml, orally taken three times daily; children aged 3 to 5 year old: 8ml, orally taken three times daily;
  Other Names: Guaifenesin, Methylephedrine and Chlorphenamine Syrup
  Arms: Injection and medications
Drug: Ibuprofen Suspension — taken under prescription
  Other Names: Motrin
  Arms: Injection and medications
Drug: salbutamol — taken under prescription
  Other Names: β2-agonists
  Arms: Injection and medications

SUMMARY:
The purpose of this study is to evaluate the effectiveness of traditional Chinese medicine for treatment of pediatric pneumonia. It is a multicenter randomized controlled trial.

DETAILED DESCRIPTION:
The retrospective case study has been finished at the National clinical research base of traditional Chinese medicine for major disease pediatric pneumonia, and the research center organized the field training of prospective-study to coordinated units. Based on the primary statistical outcomes of retrospective case study and the discussion around prospective-study during the training, investigators found it difficult to include simplex viral infection, therefore, investigators revised the inclusion criteria and treatment protocol of the pragmatic randomized controlled trial.

The block randomization is used in this trial. Random numbers are generated by SPSS software. Statistical analysis staff and those who perform the follow-up are blinded. Sample size calculation was performed, which was 369, and considering drop-out or withdrawal, investigators plan to enroll 450 patients (300 in experimental group, 150 in control).

ELIGIBILITY:
Inclusion Criteria:

* children, aged 6 months to 59 months old, diagnosed as pneumonia according to western medicine diagnostic criteria;
* diagnosed as TCM pneumonia with gasp-cough, meeting wind-heat blocking lungs pattern (feng re bi fei zheng), and phlegm-heat blocking lungs pattern (tan re bi fei zheng);
* disease progression within 72 hours;
* those whose guardians understood and assigned the informed consent;

Exclusion Criteria:

* emergency pneumonia;
* complicated with other Pulmonary Disorders attack other than pneumonia;
* complicated with primary disease of heart (congenital heart disease, myocarditis, et al), liver (ALT, and AST ≥ 1.5 times of normal value ceiling), kidney (BUN > 8.2mmol/L, or serum CR > 104 µmol/L, et al) and blood system (anemia), and those with psychopathy;
* allergic to interventional medications;
* those who are participating or have participated in other clinical trials in 3 months.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 451 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cured rate | Every day since receiving treatment, all together 10 days (times)
  Clinical symptoms and signs totally disappear, the period of lab tests return to normal is recorded.
Effectiveness time window | Every day since receiving treatment, all together 10 days (times)
  days range from treatment is received to the effectiveness is observed, and symptoms disappear

SECONDARY OUTCOMES:
TCM syndrome scores and effective rate | 10 days
  Total effective rate according to TCM syndrome differentiation and treatment, and single syndrome effective rate
Effect in fever, cough, phlegm and gasp | 10 days
  temperature, fever frequency, fever lasting time, Ibuprofen Suspension dosing; cough severity; phlegm amount, color and nature; gasp frequency, severity, all to be measured
Time of lung rales disappear completely | 10 days
  days are counted since receiving treatment, when the chest radiograph returns to normal
Check-out time | 10 days
  days counted when the patient checks out
Pulmonary disease incidence | 30 days
  unresolved pneumonia, chronic cough, cough variant asthma incidence in the follow-up

OTHER OUTCOMES:
Direct medical cost | observed during treatment in 10 days
  Medical cost including hospital expenses, examine fee, medication fee, et al, related to treatment in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng Wang, Ph.D., Study Director — Affiliated Hospital of Liaoning University of TCM; Zhenqi Wu, Principal Investigator — Affiliated Hospital of Liaoning University of TCM
Locations (6):
- China (6):
  - Affiliated Children's Hospital of Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Guangzhou Children's Hospital, Guangzhou, Guangdong
  - Affiliated Children's Hospital of Dalian Medical University, Dalian, Liaoning
  - Affiliated Hospital of Liaoning University of TCM, Shenyang, Liaoning
  - Affiliated Hospital of Shandong University of TCM, Ji'nan, Shandong
  - Affiliated Longhua Hospital of Shanghai University of TCM, Shanghai, Shanghai Municipality